CLINICAL TRIAL: NCT01190423
Title: Family-Based Treatment for Weight Restoration in Young Adults With Anorexia Nervosa
Brief Title: Treatment for Young Adults With Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20550; R34MH083914-01 (NIH)
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Anorexia Nervosa
Keywords: AN
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Family Based therapy for young adults (Experimental)
  Interventions: Behavioral: Family Based Therapy for young adults

INTERVENTIONS:
Behavioral: Family Based Therapy for young adults — Individual and Group Therapy Sessions
  Other Names: FBT; FBT-Y

SUMMARY:
Temple University is conducting a National Institute of Health funded research study designed to develop and refine a family-based treatment manual for young adults with Anorexia Nervosa as well as assess the feasibility of this out-patient psychotherapy.

DETAILED DESCRIPTION:
Anorexia Nervosa (AN) is a serious psychiatric illness that occurs in an estimated 0.5 to 3.7% of women. The illness severely affects physical, emotional, and social functioning. The mortality rates associated with this severely disabling condition are higher than those for any other psychiatric disorder and substantially higher than those expected in the general population. Lower weight at presentation, longer illness duration, and alcohol abuse are associated with a higher risk of mortality.

Treatment-outcome for adult AN is poor with a quarter of adults with AN having poor outcome. In AN, promising outcomes are seen in family-based treatment (FBT) for adolescent patients who present between the ages of 12 to 18 with a short duration of illness. A manualized version of FBT has now been tested in several studies and case series, showing that well over 80% of participants had good or intermediate outcome at post-treatment. Despite its efficacy with adolescents, FBT has not been utilized with young adults.

The purpose of this study is to develop and refine FBT to promote weight gain in young adults with Anorexia Nervosa.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV criteria for AN (restricting/binge-purge type) (BMI 16.0-18.5)
* Medically stable for outpatient treatment
* Availability of at least one supportive adult of choice in study client's environment
* Stable dose of psychotropic medication (8 weeks) for co-morbid condition

Exclusion Criteria:

* Associated physical illness that necessitates hospitalization
* Psychotic illness or other mental illness requiring hospitalization
* Current dependence on drugs or alcohol
* Physical conditions (e.g. diabetes mellitus, pregnancy) known to influence eating or weight
* Previous Family-Based Treatment for Anorexia

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2010-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Weight (BMI) | 6 months of treatment

SECONDARY OUTCOMES:
Changes in shape and weight concerns as measured with Eating Disorder Examination subscales | 18 therapy sessions or 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Eunice Y Chen, PhD, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Chen EY, Weissman JA, Zeffiro TA, Yiu A, Eneva KT, Arlt JM, Swantek MJ. Family-Based Therapy for Young Adults with Anorexia Nervosa Restores Weight. Int J Eat Disord. 2016 Jul;49(7):701-7. doi: 10.1002/eat.22513. Epub 2016 Apr 1. PMID 27037965
- See also: For More Information About The Study — http://sites.temple.edu/tedp